CLINICAL TRIAL: NCT06534099
Title: Effect of Wuqinxi on the Balance Ability of Older Women With a History of Falls: A Randomized Controlled Trial
Brief Title: Balance Ability of Older Women With a History of Falls
Acronym: Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cheng Liang (Other)
Responsible Party: Sponsor-Investigator, Cheng Liang, Principal Investigator, Chengdu Sport University
Organization: Chengdu Sport University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Sichuan Fitness Qigong Center; Sichuan Fitness Qigong Center (Other: Chengdu Sport University)
Record Dates: First submitted 2024-07-29; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Falls
Keywords: older Women; Falls
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Without changing their original lifestyle habits, weekly follow-ups were conducted by the experimenters via telephone or face-to-face interviews to ensure that the participants did not engage in other forms of regular fitness activities.
  Interventions: Other: Control
- Experimental (Experimental): The Wuqinxi exercise regimen was conducted under the guidance of a professional Wuqinxi instructor, where the experimental group practiced the five animal forms of the exercise, which include the Tiger, Deer, Bear, Ape, and Bird forms. The exercise period was 24 weeks, with the first 4 weeks designated as the learning phase and weeks 5 to 24 as the consolidation and reinforcement phase. The frequency of exercise was three times per week, with each session lasting 70 minutes, including 10 minutes for warm-up and relaxation activities.
  Interventions: Other: Control; Other: Experimental

INTERVENTIONS:
Other: Control — Without changing their original lifestyle habits, weekly follow-ups were conducted by the experimenters via telephone or face-to-face interviews to ensure that the participants did not engage in other forms of regular fitness activities.
  Other Names: Control Group
Other: Experimental — The Wuqinxi exercise regimen was conducted under the guidance of a professional Wuqinxi instructor, where the experimental group practiced the five animal forms of the exercise, which include the Tiger, Deer, Bear, Ape, and Bird forms. The exercise period was 24 weeks, with the first 4 weeks designated as the learning phase and weeks 5 to 24 as the consolidation and reinforcement phase. The frequency of exercise was three times per week, with each session lasting 70 minutes, including 10 minutes for warm-up and relaxation activities.
  Other Names: Experimental group
  Arms: Experimental

SUMMARY:
This study aims to investigate the effects of regular practice of Chinese fitness Qigong, Wuqinxi, on the balance ability of older women with a history of falls. Participants in the experimental group (n=35) and the control group (n=36), matched for age, height, and weight, were included in the study. The experimental group underwent a 24-week (3 times per week, 70 minutes per session) Wuqinxi exercise regimen. Changes in dynamic and static balance abilities of the participants were tested at weeks 0, 12, and 24. A 24-week Wuqinxi exercise regimen increased the static and dynamic balance abilities in both directions for older women with a history of falls. Compared to 12 weeks, a longer Wuqinxi exercise regimen further enhanced the static balance ability in the open-eye state.

DETAILED DESCRIPTION:
The Wuqinxi exercise regimen was conducted under the guidance of a professional Wuqinxi instructor, where the experimental group practiced the five animal forms of the exercise, which include the Tiger, Deer, Bear, Ape, and Bird forms. The exercise period was 24 weeks, with the first 4 weeks designated as the learning phase and weeks 5 to 24 as the consolidation and reinforcement phase. The frequency of exercise was three times per week, with each session lasting 70 minutes, including 10 minutes for warm-up and relaxation activities. Participants practiced to fixed voice prompts and musical rhythms, completing four full sets of Wuqinxi movements, each set taking approximately 14 minutes with a 1-minute interval in between. Following the research design of Cheng et al, after completing each set of movements, participants immediately pressed on the radial artery to test the pulse beats for 10 seconds and reported their heart rate per minute to the experimenters. The exercise intensity was controlled within the range of (220 - age) x (55% to 65%). Participants were allowed to take a break if their heart rate was too high. Additionally, without changing their original lifestyle habits, weekly follow-ups were conducted by the experimenters via telephone or face-to-face interviews to ensure that the participants did not engage in other forms of regular fitness activities.

Compliance with the exercise regimen was managed through the following methods: regular supervision, with professional staff overseeing the training to ensure participants followed the set plan; completion of training logs, requiring participants to record detailed information about each training session, including content, duration, and intensity; and regular follow-ups, maintaining contact with participants through phone calls, WeChat, or face-to-face meetings to understand their training status and provide necessary support.

The balance ability tests were conducted on three occasions: at baseline, at the 12th week, and at the 24th week. The Good Balance balance testing device, manufactured in Finland, was used for all participants, which has been demonstrated to have good reliability and validity. Both static and dynamic balance tests were conducted with participants standing on the test platform using a stopwatch to measure the time that participants could stand on one leg with eyes open and closed.

ELIGIBILITY:
Inclusion criteria:

* Female, aged between 60 and 70 years
* At least one accidental fall within the past year
* Undergone a physical examination for cardiac function
* Have the intention to exercise and are able to complete the entire experimental process
* In compliance with the Declaration of Helsinki and have signed an informed consent form.

Exclusion criteria:

* Regular exercise habits through other means within the past 6 months
* Foot deformity, abnormal gait
* A history of severe lower limb trauma
* Epilepsy, motor disorders
* Cardiovascular diseases.

Ages: 60 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-05 (Actual)

PRIMARY OUTCOMES:
Balance Ability Testing | 24 weeks
  The balance ability tests were conducted on three occasions: at baseline, at the 12th week, and at the 24th week. The Good Balance balance testing device, manufactured in Finland, was used for all participants, which has been demonstrated to have good reliability and validity. Both static and dynamic balance tests were conducted with participants standing on the test platform using a stopwatch to measure the time that participants could stand on one leg with eyes open and closed.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Yi, Dr, Principal Investigator — Chengdu Sport University
Locations (1):
- Chengdu Sport University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No